CLINICAL TRIAL: NCT06271382
Title: The Effect Of Acupressure and Foot Exercise on Ankle Brachial Index in Individuals With Type 2 Diabetes: A Randomized Controlled Trial
Brief Title: The Effect Of Acupressure and Foot Exercise on Ankle Brachial Index in Individuals With Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Saadet Can Çiçek, Associate Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AIBU-SBF-SA-05
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Acupressure; Ankle Brachial Index; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupressure Group (Experimental): In the research, acupressure will be applied to the patients in the acupressure group on LR 3 Taichung(LR 3), Tai Xi (KI 3), San Yin Jiao(SP 6), Xue Hai (SP 10), Zusanli(ST 36 ) points.
  Interventions: Other: Acupressure Group
- Sham Acupressure Group (Sham Comparator): The same process will continue with the acupressure group by applying pressure to different points in the group where acupressure is applied to the sham points.
  Pressure will be applied on the bone area where the meridians do not pass, parallel to the points where acupressure is applied to the sham points (approximately 1-1.5 cm away).
  Interventions: Other: Sham Acupressure Group
- Foot Ankle Exercise Group (Experimental): The foot and ankle exercise complex includes the following exercises.
  1. Pulling the foot towards itself from the ankle up
  2. Bending the foot downwards from the ankle
  3. Opening the feet like a fan, moving the toes inward and outward, left and right
  4. Circling exercise with ankle
  5. Towel folding exercise
  6. Bottle rolling exercise under your feet (The water in the bottle will be warm tap water)
  Interventions: Other: Foot Ankle Exercise Group

INTERVENTIONS:
Other: Acupressure Group — In the research, the participant in the acupressure group will receive acupressure application 3 times a week for 2 weeks, a total of 6 times.
  Depending on the preparation and pressure time on the 5 selected points (a total of 10 points will be applied since the partner of each point on the other extremity will be applied), the session duration for an individual will be approximately 18-20 minutes.
  Arms: Acupressure Group
Other: Sham Acupressure Group — Depending on the preparation and pressure time on the 5 selected sham points (a total of 10 points will be applied since the partner of each point on the other extremity will be applied), the session duration for an individual will be approximately 18-20 minutes.
  Patients in the sham acupressure group will receive acupressure 6 times in total, 3 times a week for 2 weeks. The practitioner will do the first acupressure at the Family Health Center, and the person with type 2 diabetes will do the others at home. Ankle Brachial Index evaluation will be performed by the researcher at the Family Health Center a total of 3 times before the intervention, 1 week after the intervention and 2 weeks after the intervention.
  Arms: Sham Acupressure Group
Other: Foot Ankle Exercise Group — Exercise will be performed regularly for 2 weeks, 3 days a week for a maximum of 30 minutes.
  Arms: Foot Ankle Exercise Group

SUMMARY:
This study was planned with a randomized controlled experimental design to examine the effects of acupressure and ankle exercises on ankle brachial index in individuals with Type 2 diabetes.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) is a health problem that affects many lifelong systems and organs throughout the world, increases the risk of premature death, affects the individual, family, society and the world, has a serious spiritual and financial care burden, and has important and vital consequences.

Diabetes can cause damage to nerves as well as small and large vessels. Patients who have had DM for a long time will experience circulatory disorders in the upper and lower extremities.

Ankle-Brachial Index (ABI) is a non-invasive examination of blood vessels that functions to detect clinical signs and symptoms of ischemia, reduced peripheral perfusion that can lead to angiopathy and diabetic neuropathy.

Studies indicate that foot exercise and acupressure application can be used as an alternative intervention to increase the value of the ankle-brachial index in patients with type 2 diabetes.

When the literature was examined, no comprehensive study could be found comparing the effect of foot exercise and acupressure application on the Ankle Brachial Index in diabetic patients in our country. It is thought that acupressure application and ankle exercises will accelerate peripheral circulation and may be effective on the ankle brachial index.

This study was planned with a randomized controlled experimental design to examine the effects of acupressure and ankle exercises on ankle brachial index in individuals with Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with type 2 diabetes
* Be 18 years or older
* Ability to speak Turkish
* Ability to establish verbal communication
* Volunteering to participate in the research

Exclusion Criteria:

* Presence of any psychiatric disease diagnosed by a physician
* Presence of diabetic ulcers on both feet and legs
* Presence of any amputation in the foot or leg
* Having myalgia in the foot,
* Foot fracture
* Edema in the feet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-04-24 (Estimated); Study Completion 2025-04-24 (Estimated)

PRIMARY OUTCOMES:
Ankle Brachial Index | 2 week
  The ABI evaluation form includes right and left ankle blood pressure values, right and left arm blood pressure values and the ratios of these values.
  ABI interpretation:
  0.9-1.3 is normal, 0.8-0.9 Risky or Mild Stenosis, 0.8-0.4 Moderate Stenosis, <0.4 Severe Stenosis

CONTACTS AND LOCATIONS:
Overall Officials: Saadet CAN ÇİÇEK, Study Director — http://www.ibu.edu.tr/tr
Locations (1):
- Beşkavaklar Aile Sağlığı Merkezi, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No